CLINICAL TRIAL: NCT00411463
Title: Psychotherapy for Bipolar II Depression, Pilot Study, Phase II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Holly Swartz, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0608080
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Bipolar II Disorder
Keywords: Interpersonal Therapy; Social Rhythm Therapy; Bipolar Disorder; Depression; Seroquel
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychotherapy (Experimental): Subjects randomized to the Psychotherapy arm will receive Interpersonal and Social Rhythm Therapy (IPSRT-BPII)
  Interventions: Behavioral: Interpersonal and Social Rhythm Therapy (IPSRT-BPII)
- Medication (Experimental): Subjects randomized to the medication arm will receive the FDA approved medication Seroquel (quetiapine)
  Interventions: Drug: Seroquel

INTERVENTIONS:
Behavioral: Interpersonal and Social Rhythm Therapy (IPSRT-BPII) — IPSRT is comprised of three components: psychoeducation, social rhythm therapy, and standard IPT as developed for unipolar depression.
  Psychoeducation focuses on a) the illness and its consequences, b) treatment options and associated side effects, and c) prodromal symptoms/detection of early warning symptoms.
  Other Names: IPSRT
  Arms: Psychotherapy
Drug: Seroquel — Subjects will be started at 100 mg/day titrated to a maximum of 800 mg /day
  Day 1-BID doses totaling 100 mg/day, increased to 400 mg/day on Day 4 in increments of up to 100 mg/day in BID divided doses, by Day 6 begin titration up to a maximum dose of 800 mg/day in increments no greater than 200 mg/day.
  This titration schedule may be adjusted based on the subject's response and ability to tolerate Seroquel.
  Subjects who are unable to tolerate the study medications, or for whom the study medications are an inappropriate clinical choice, will be treated openly by a clinic physician according to the standard of care guidelines designated by the American Psychiatric Association (2002) for the treatment of bipolar disorder.
  Other Names: Quetiapine
  Arms: Medication

SUMMARY:
Purpose of this study is to examine the effectiveness of an experimental psychotherapy (talk therapy) for the treatment of bipolar II depression. The name of this psychotherapy is Interpersonal and Social Rhythm Therapy for Bipolar II Depression (IPSRT-BPII). Subjects will be randomly assigned to receive either IPSRT-BPII or the medication Seroquel (quetiapine) to manage their symptoms of bipolar II depression. Subjects will receive the assigned therapy for up to 20 weeks.

DETAILED DESCRIPTION:
The proposed pilot study is an experimental design intended to investigate the preliminary efficacy of Interpersonal Social Rhythm Therapy for Bipolar II Depression (IPSRT-BPII). A total of 56 eligible subjects with a diagnosis of bipolar II disorder will be randomly assigned to one of two treatment groups : Seroquel (n=28) or IPSRT-BPII (n=28). Following baseline assessment, all participants will undergo up to 20 weeks of their assigned treatment. Patients assigned to IPSRT-BPII who fail to respond (at least 50% reduction in HRSD-25 scores and YMRS ≤ 10) by week 12 will have Seroquel added to IPSRT-BPII. Subjects who achieve remission (defined as 3 consecutive weeks where both HRSD-25 and YMRS scores average ≤ 7) and have participated in the trial for a minimum of 12 weeks will be moved into a continuation phase where they will receive maintenance treatment (bi-monthly therapy sessions and/or pharmacotherapy) until week 20. Patients who do not achieve remission by Week 20 will be discontinued from treatment and referred for follow-up care. All subjects (remitters and non-remitters) will be assessed at 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV Criteria for Bipolar Disorder, Type II, currently depressed;
2. HRSD-25 ≥15
3. Age 18-65 years;
4. Able to give informed consent;
5. Women of child bearing potential will be included if they agree to use adequate contraception for the duration of the study.

Exclusion Criteria:

1. Not competent to give informed consent in the opinion of the investigator (e.g., psychotic at time of evaluation);
2. Unwilling or unable to comply with study requirements;
3. Meets DSM-IV criteria for borderline personality disorder or antisocial personality disorder;
4. Active substance abuse within the past 6 months(episodic abuse related to mood episodes will not exclude a subject);
5. Currently a high suicide risk, as assessed by an active plan and intent to behave in a way that risks ending ones life;
6. Non-English speaking;
7. Significant, unstable, medical illness that might confound symptom scores or preclude treatment with pharmacotherapy
8. Currently applying for disability because of psychiatric illness (we have found that these individuals have a vested interested in appearing to remain ill which potentially confounds outcome scores).
9. Women who are pregnant, lactating or plan to become pregnant during their study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Swartz, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh /University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Swartz HA, Frank E, Cheng Y. A randomized pilot study of psychotherapy and quetiapine for the acute treatment of bipolar II depression. Bipolar Disord. 2012 Mar;14(2):211-6. doi: 10.1111/j.1399-5618.2012.00988.x. PMID 22420597

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychotherapy: Subjects randomized to the Psychotherapy arm will receive Interpersonal and Social Rhythm Therapy (IPSRT-BPII)
  Interpersonal and Social Rhythm Therapy (IPSRT-BPII): IPSRT is comprised of three components: psychoeducation, social rhythm therapy, and standard IPT as developed for unipolar depression.
  Psychoeducation focuses on a) the illness and its consequences, b) treatment options and associated side effects, and c) prodromal symptoms/detection of early warning symptoms.
- Medication: Subjects randomized to the medication arm will receive the FDA approved medication Seroquel (quetiapine)
  Seroquel: Subjects will be started at 100 mg/day titrated to a maximum of 800 mg /day
  Day 1-BID doses totaling 100 mg/day, increased to 400 mg/day on Day 4 in increments of up to 100 mg/day in BID divided doses, by Day 6 begin titration up to a maximum dose of 800 mg/day in increments no greater than 200 mg/day.
  This titration schedule may be adjusted based on the subject's response and ability to tolerate Seroquel.
  Subjects who are unable to tolerate the study medications, or for whom the study medications are an inappropriate clinical choice, will be treated openly by a clinic physician according to the standard of care guidelines designated by the American Psychiatric Association (2002) for the treatment of bipolar disorder. Subjects receiving standard of care treatment will continue to be seen and assessed per the protocol schedule.
Period: Overall Study
Arm/Group | Psychotherapy | Medication
Started | 14 | 11
Completed | 11 | 8
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychotherapy | Medication | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.7) | 32.1 (12.8) | 36.1 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Greater Than or Equal to 50% Reduction in Depression Scores, With a Mania Score Less Than or Equal to 10
Description: Overall response rates (defined as greater than or equal to 50% reduction in depression scores without an increase in mania scores) were 29% (n=4) in the IPSRT group and 27% (n=3) in the quetiapine group. HRSD-25 scores are based on first 17 responses. Eight items are scored on a 5-pt scale, from 0 (not present) to 4 (severe.) Other nine items on the assessment are scored from 0-2. The higher the score on the HRSD-25, the worse the outcome is considered to be. A score of 0-7 is considered to be normal; 8-13 indicates mild depression, 14-18 indicates moderate depression, 19-22 indicates severe depression, and any score greater than or equal to 23 indicates very severe depression. The YMRS is an 11 point assessment. There are 4 items assessed on a scale ranging from 0 to 8 and the other 7 items are graded on a 0 to 4 scale. As with the HRSD, the higher the score on the YMRS indicates the presence of more or more severe manic symptoms and is associated with a worse outcome.
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Psychotherapy | Medication
Number analyzed (Participants) | 14 | 11
participants
  50% reduction in HRSD 25 score and YMRS <= 10 | 4 | 3
  Non-responder | 10 | 8

2. Secondary Outcome: Quality of Life (QOL) Collected Using the Q-LES-Q (Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form)
Description: The total score is derived by summing item scores 1 to 14. Higher scores are indicative of greater enjoyment or satisfaction in each domain. The Q-LES-Q-SF % maximum total score is calculated as 100% × (Q-LES-Q-SF total score - 14) / 56, and can range from 0% to 100%.
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on Q-LES-Q scale
Groups:
- Psychotherapy: Patients assigned to talk therapy (IPSRT) intervention during 12 weeks of active enrollment in study.
- Medication: Patients taking Quetiapine (Seroquel) during 12 weeks of active treatment.
Arm/Group | Psychotherapy | Medication
Number analyzed (Participants) | 14 | 11
scores on Q-LES-Q scale
  Baseline | 34.6 [30.0 to 39.3] | 40.0 [35.2 to 45.6]
  Post-Intervention | 37.0 [32.0 to 41.9] | 48.7 [43.2 to 54.3]

3. Secondary Outcome: Descriptive Measures of the Feasibility of IPSRT-BPII
Description: Feasibility was assessed by ability to enroll, randomize, and retain participants in this trial. Completion of the study was used as evidence of feasibility.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total number of participants
Arm/Group | Psychotherapy | Medication | Total
Number analyzed (Participants) | 14 | 11 | 25
Participants | 11 | 8 | 19

4. Secondary Outcome: Number of Participants With a Response
Description: Number of participants with response defined as an average of 50% (or greater) reduction in the subject's baseline HRSD-25 score over three consecutive weeks and a current YMRS score ≤ 10
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Psychotherapy | Medication
Number analyzed (Participants) | 14 | 11
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Psychotherapy | Medication
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No